CLINICAL TRIAL: NCT02231619
Title: The Feasibility of Replacing In-person Follow-up for Early Medical Abortion With a Low Sensitivity Pregnancy Test, Symptom Checklist and Text Messages in the South African Public Sector Setting.
Brief Title: Use of Low Sensitivity Pregnancy Test for Self-assessment of Medical Abortion
Acronym: m-Assist+
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cape Town (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Deborah Constant, Ms, University of Cape Town
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 677/2013
Record Dates: First submitted 2014-08-31; First posted 2014-09-04 (Estimated); Last update posted 2015-11-09 (Estimated); Status verified 2015-11

CONDITIONS: Completion of Medical Abortion
Keywords: feasibility; self assessment; medical abortion; low sensitivity urine pregnancy test; South Africa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Demonstration of LSUPT at baseline (No Intervention): This group conduct a LSUPT on their own urine sample at baseline with assistance from a fieldworker.
- Baseline verbal instruction of LSUPT (Active Comparator): Verbal instruction on how to do LSUPT at baseline
  Interventions: Behavioral: Baseline verbal instruction on LSUPT

INTERVENTIONS:
Behavioral: Baseline verbal instruction on LSUPT
  Other Names: Low sensitivity urine pregnancy test
  Arms: Baseline verbal instruction of LSUPT

SUMMARY:
The purpose of the study is to design a self-assessment package that could be the preferred option to a follow-up visit at the clinic by the majority of women having early medical abortion.

ELIGIBILITY:
Inclusion Criteria:

1. Already be signed up to do a medical abortion at this clinic
2. Be willing to come to all clinic appointments and be accessible by phone for 2 weeks after sign up for the study
3. Own a cellphone to which will be sent medical abortion-related information and messaging.

Exclusion Criteria:

1. Be doing a medical abortion due to failed natural miscarriage 2. Not have a working cellphone

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 525 (Actual)
Dates: Start 2014-08; Primary Completion 2015-08 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Accurate self-assessment of medical abortion using a low sensitivity pregnancy test | 12 months
  Participants will be randomized to 2 groups. Women in Group A will conduct a baseline low sensitivity urine pregnancy test (LSUPT) on their own urine specimen at their clinic visit with help from the fieldworker. Group B will receive a standardized set of verbal instructions on how to do the test. Both groups will do a LSUPT at home on Day 12.

CONTACTS AND LOCATIONS:
Locations (1):
- Nolungile Youth Clinic, Khayelitsha, Cape Town, Western Province, South Africa

REFERENCES:
- [Derived] Constant D, Harries J, Daskilewicz K, Myer L, Gemzell-Danielsson K. Is self-assessment of medical abortion using a low-sensitivity pregnancy test combined with a checklist and phone text messages feasible in South African primary healthcare settings? A randomized trial. PLoS One. 2017 Jun 22;12(6):e0179600. doi: 10.1371/journal.pone.0179600. eCollection 2017. PMID 28640845